CLINICAL TRIAL: NCT00003084
Title: A Randomized Phase II Trial of Taxol/VP-16/Estramustine vs. Ketoconazole/Doxorubicin/Vinblastine/Estramustine in Androgen Independent Prostate Cancer
Brief Title: Combination Chemotherapy With Ketoconazole in Treating Patients With Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DM97-022; P30CA016672 (NIH); MDA-DM-97022 (Other: UT MD Anderson Cancer Center); NCI-T97-0023; CDR0000065783 (Registry Identifier: NCI PDQ)
Record Dates: First submitted 1999-11-01; First posted 2004-05-24 (Estimated); Last update posted 2012-07-30 (Estimated); Status verified 2012-07

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; stage I prostate cancer; stage II prostate cancer; stage III prostate cancer; stage IV prostate cancer; recurrent prostate cancer; Chemotherapy; Ketoconazole; Estramustine; Etoposide; Paclitaxel; Doxorubicin; Vinblastine
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Doxorubicin; Estramustine; Etoposide; Ketoconazole; Paclitaxel; Vinblastine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm I (Estramustine + Etoposide) (Experimental): Arm I: Oral Estramustine 3 x day + oral Etoposide 2 x day on days 1-14 + Paclitaxel IV over 1 hour Day 2, repeats every 21 days.
  Interventions: Drug: Estramustine phosphate sodium; Drug: Etoposide; Drug: Paclitaxel
- Arm II (Chemotherapy + Ketoconazole) (Experimental): Arm II: Doxorubicin IV Days 1, 15, and 29, Vinblastine IV Days 8, 22, and 36, Oral Ketoconazole 3 x day on Days 1-7, 15-21, + 29-35, and Oral Estramustine 3 x day on Days 8-14, 22-28, and 36-42; 6 weeks of alternating chemotherapy and 2 weeks rest, for 8 week course.
  Interventions: Drug: Doxorubicin Hydrochloride; Drug: Estramustine phosphate sodium; Drug: Ketoconazole; Drug: Vinblastine

INTERVENTIONS:
Drug: Doxorubicin Hydrochloride — Doxorubicin IV on days 1, 15, and 29.
  Other Names: Adriamycin; Rubex
  Arms: Arm II (Chemotherapy + Ketoconazole)
Drug: Estramustine phosphate sodium — Arm I: Oral estramustine three times a day for 21 day cycle.
  Arm II: Oral estramustine three times a day on days 8-14, 22-28, and 36-42 in 8 week cycle.
  Other Names: Emcyt
Drug: Etoposide — Oral etoposide twice daily on days 1-14.
  Other Names: VePeside
  Arms: Arm I (Estramustine + Etoposide)
Drug: Ketoconazole — Oral ketoconazole three times a day on days 1-7, 15-21, and 29-35.
  Other Names: Nizoral
  Arms: Arm II (Chemotherapy + Ketoconazole)
Drug: Paclitaxel — IV over 1 hour on day 2.
  Other Names: Taxol
  Arms: Arm I (Estramustine + Etoposide)
Drug: Vinblastine — IV on days 8, 22, and 36.
  Other Names: Velban
  Arms: Arm II (Chemotherapy + Ketoconazole)

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Randomized phase II trial to study the effectiveness of combination chemotherapy consisting of paclitaxel, etoposide, and estramustine as compared with ketoconazole plus doxorubicin, vinblastine, and estramustine in treating patients with prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the clinical benefit of two combination chemotherapy regimens, paclitaxel, etoposide, and estramustine vs ketoconazole, doxorubicin, vinblastine, and estramustine in patients with androgen independent prostate cancer, as measured by prostate specific antigen (PSA)-based response rate, time to progression, and overall survival. II. Identify the most promising regimen to use in a phase III trial based on toxic effects, PSA-based response rates, and clinical benefit.

OUTLINE: This is a randomized multicenter study. Patients are stratified according to risk group: low volume disease (no more than 2 lesions on bone scan), intermediate volume (more than 2 bone lesions confined to axial skeleton), or high volume (bone lesions in appendicular skeletal or visceral lesions). Patients are randomized to one of two treatment arms. Arm I: Patients receive oral estramustine three times a day and oral etoposide twice daily on days 1-14 and paclitaxel IV over 1 hour on day 2. Treatment repeats every 21 days. Arm II: Patients receive doxorubicin IV on days 1, 15, and 29, vinblastine IV on days 8, 22, and 36, oral ketoconazole three times a day on days 1-7, 15-21, and 29-35, and oral estramustine three times a day on days 8-14, 22-28, and 36-42. This regimen consists of 6 weeks of alternating chemotherapy and 2 weeks rest, for an 8 week course. Treatment continues in the absence of disease progression or unacceptable toxicity.

PROJECTED ACCRUAL: A total of 92 patients (46 per treatment arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed adenocarcinoma of the prostate Androgen independent disease progression -Castrate testosterone level of less than 40 ng/dL (if medically achieved, treatment must be maintained continuously) -Prostate specific antigen (PSA) at least 4 ng/mL and rising on at least 2 consecutive measurements No variant histologies such as ductal carcinoma (endometrioid or cribiform) or small cell carcinoma Brain metastases controlled

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Zubrod 0-3 Life expectancy: At least 12 weeks Hematopoietic: Absolute neutrophil count at least 1500/mm3 Platelet count at least 100,000/mm3 Hemoglobin greater than 9.5 g/dL (without transfusion support) Hepatic: Bilirubin and transaminase less than 2 times the upper limit of normal Renal: Creatinine no greater than 2.0 mg/dL OR Estimated creatinine clearance at least 35 mL/min Cardiovascular: No clinical history of heart disease Normal ECG OR Ejection fraction (ECHO, MUGA, or ventriculography) at least 45% Other: Spinal cord compression controlled No active peptic ulcer disease No active, or likely to become active, second malignancy

PRIOR CONCURRENT THERAPY: Biologic therapy: No prior ketoconazole Chemotherapy: No prior doxorubicin, vinblastine, estramustine, paclitaxel, or etoposide No greater than one prior cytotoxic therapy No other concurrent chemotherapy At least 8 weeks since prior mitomycin At least 60 days since prior suramin Endocrine therapy: No antiandrogen therapy such as flutamide or nilutamide within 4 weeks (6 weeks for bicalutamide) without response OR Progression since antiandrogen withdrawal Prior dexamethasone therapy discontinued Radiotherapy: At least 10 weeks since prior strontium Sr 89 and no more than 1 prior regimen No concurrent strontium Sr 89 Surgery: Not specified Other: No other concurrent therapy for prostate cancer No concurrent H2 blockers, omeprazole, or antacids No concurrent terfenadine and astemizole

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 1997-12; Primary Completion 2002-11 (Actual); Study Completion 2002-11 (Actual)

PRIMARY OUTCOMES:
Prostate specific antigen (PSA)- based Response Rate | 8 week cycle

CONTACTS AND LOCATIONS:
Overall Officials: Randall E. Millikan, MD, PhD, Study Chair — M.D. Anderson Cancer Center
Locations (1):
- University of Texas - MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Result] Millikan R, Thall PF, Lee SJ, Jones D, Cannon MW, Kuebler JP, Wade J 3rd, Logothetis CJ. Randomized, multicenter, phase II trial of two multicomponent regimens in androgen-independent prostate cancer. J Clin Oncol. 2003 Mar 1;21(5):878-83. doi: 10.1200/JCO.2003.04.057. PMID 12610188
- See also: UT MD Anderson Cancer Center Website — http://www.mdanderson.org